CLINICAL TRIAL: NCT04766996
Title: PROUD Study - Preventing Opioid Use Disorders
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Loss of surgery team member deemed the study procedures impossible to achieve, and no replacement could be found in a timely manner to complete trial as initially planned.
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Kelly Wiltse Nicely, Assistant Professor, Emory University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00002021
Record Dates: First submitted 2021-02-19; First posted 2021-02-23 (Actual); Results first posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Anesthesia; Opioid Use
Keywords: Hip replacement; Opioid free; Perioperative period; Team work
MeSH Terms: interventions — Acetaminophen; Pregabalin; Prednisone; Meloxicam; Omeprazole; Tramadol; Diclofenac; Ondansetron; Famotidine; Metoclopramide; Midazolam; Lidocaine; Propofol; Cefazolin; Tranexamic Acid; Calcium Dobesilate; Bupivacaine; Ketorolac Tromethamine

STUDY DESIGN:
Intervention Model Description: Matched Prospective Case with Retrospective Control Study and Staff Survey
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Prospective cases undergoing non-opioid drug regimen (Experimental): Prospective study participants undergoing unilateral total hip replacement surgery and non-opioid drug regimen perioperatively
  Interventions: Behavioral: Guided mindfulness exercises; Other: Self-administered aromatherapy; Drug: Baby aspirin; Drug: Tylenol/Acetaminophen; Drug: Pregabalin; Drug: Prednisone; Drug: Meloxicam; Drug: Prilosec; Drug: Tramadol; Drug: Voltaren; Drug: Zofran; Drug: Pepcid; Drug: Reglan; Drug: Versed; Drug: Lidocaine; Drug: Propofol; Drug: Ancef; Drug: Tranexamic Acid (TXA); Drug: Decadron; Drug: Bupivacaine hydrochloride; Drug: Toradol
- Retrospective control underwent opioid drug regimen (No Intervention): Retrospective controls that underwent unilateral total hip replacement surgery and used opioid drug regimen perioperatively
- Professional Staff (No Intervention): Staff that participate in the implementation of the opioid free surgical protocol will be completing team assessment surveys seeking their opinion about interprofessional teamwork and communication.

INTERVENTIONS:
Behavioral: Guided mindfulness exercises — Guided Meditation twice daily
  Arms: Prospective cases undergoing non-opioid drug regimen
Other: Self-administered aromatherapy — Self-administered aromatherapy every 6 hours and at bedtime
  Arms: Prospective cases undergoing non-opioid drug regimen
Drug: Baby aspirin — Baby aspirin 81mg: Twice daily for 6 weeks after surgery
  Arms: Prospective cases undergoing non-opioid drug regimen
Drug: Tylenol/Acetaminophen — Tylenol/Acetaminophen 1000mg: Pre-operative one dose; Every 8 hours for three weeks after surgery
  Arms: Prospective cases undergoing non-opioid drug regimen
Drug: Pregabalin — Pregabalin 25mg:
  Twice a day for two weeks before surgery; Pre-operative 25-100 mg; Twice a day for two weeks after surgery
  Arms: Prospective cases undergoing non-opioid drug regimen
Drug: Prednisone — Prednisone 5mg: Daily for three weeks after surgery
  Arms: Prospective cases undergoing non-opioid drug regimen
Drug: Meloxicam — Meloxicam 7.5mg:
  Twice a day, with food, for two weeks before surgery; Twice a day, with food, for two weeks after surgery
  Arms: Prospective cases undergoing non-opioid drug regimen
Drug: Prilosec — Prilosec 20mg:
  Daily for two weeks before surgery; Daily for for two weeks after surgery
  Arms: Prospective cases undergoing non-opioid drug regimen
Drug: Tramadol — Rescue pain medicine Tramadol 50mg up to three times a day as needed will be provided for rescue pain
  Arms: Prospective cases undergoing non-opioid drug regimen
Drug: Voltaren — Voltaren 1% topical arthritis gel up to 4 times daily pre-operative only
  Arms: Prospective cases undergoing non-opioid drug regimen
Drug: Zofran — Zofran 4 mg pre-operative
  Arms: Prospective cases undergoing non-opioid drug regimen
Drug: Pepcid — Pepcid 20 mg pre-operative
  Arms: Prospective cases undergoing non-opioid drug regimen
Drug: Reglan — Reglan 10 mg pre-operative
  Arms: Prospective cases undergoing non-opioid drug regimen
Drug: Versed — Versed 2 mg pre-operative
  Arms: Prospective cases undergoing non-opioid drug regimen
Drug: Lidocaine — Lidocaine (preservative free) height based dosing for subarachnoid block intraoperatively
  Arms: Prospective cases undergoing non-opioid drug regimen
Drug: Propofol — Propofol 10-125 mcg/kg/min intraoperative
  Arms: Prospective cases undergoing non-opioid drug regimen
Drug: Ancef — Ancef 2-3 gm weight-based dosing intraoperative
  Arms: Prospective cases undergoing non-opioid drug regimen
Drug: Tranexamic Acid (TXA) — Tranexamic Acid (TXA) 2 gm intraoperative
  Arms: Prospective cases undergoing non-opioid drug regimen
Drug: Decadron — Decadron 10 mg intraoperative
  Arms: Prospective cases undergoing non-opioid drug regimen
Drug: Bupivacaine hydrochloride — Local anaesthetic 0.5% bupivacaine hydrochloride intraoperative
  Arms: Prospective cases undergoing non-opioid drug regimen
Drug: Toradol — Toradol nonsteroidal anti-inflammatory drug max 30 mg intraoperative
  Arms: Prospective cases undergoing non-opioid drug regimen

SUMMARY:
The objective of this study is to pilot an opioid free anesthetic protocol for patients undergoing total hip replacement.

DETAILED DESCRIPTION:
The objective of this study is to pilot an opioid free anesthetic protocol for patients undergoing total hip replacement. The study team identified alternative pharmacologic methods to block pain pathways to reduce or even eliminate the need for opioids in the intra- and postoperative periods, with the goal of decreasing or eliminating exposure to opioids. A secondary objective is to assess two core competencies for interprofessional collaborative practice (Interprofessional Communication and Teams; and Teamwork) within the interprofessional care team implementing the opioid free protocol.

ELIGIBILITY:
Inclusion Criteria Intervention group:

* Prospective study participants undergoing unilateral total hip replacement surgery between the months of February through May, 2021

Inclusion Criteria Control:

* Retrospective controls selected from the Emory Healthcare System Clinical Data Warehouse that underwent unilateral total hip replacement surgery between the months of February through May, 2020

Inclusion Criteria Professional Staff:

* All staff that participate in the implementation of the opioid free surgical protocol.

Exclusion Criteria:

* Participants that do not speak English will not be eligible for participation in the study.
* Individuals less than 18 years of age will not be included for participation in the study.
* Individuals with cognitive impairment or the inability to provide informed consent will not be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2021-12-27 (Actual); Study Completion 2021-12-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wiltse Nicely, PhD, CRNA, Principal Investigator — Emory University
Locations (1):
- Emory University Orthopaedic and Spine Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in peer reviewed publication(s) will be shared after de-identification.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available for sharing beginning 6 months and ending 36 months following article publication.
Access Criteria: Data will be available for sharing with investigators whose proposed use of the data have been approved by an independent review committee identified for that purpose. Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in Emory University's data warehouse but without investigator support other than deposited metadata. Information regarding the Emory Dataverse can be found at: http://sco.library.emory.edu/dataverse/index.html
URL: http://sco.library.emory.edu/dataverse/index.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Emory Orthopaedics & Spine Center in Atlanta, Georgia, USA. Participant enrollment began May 17, 2021 and the final follow-up assessment occurred December 27, 2021.
Groups:
- Prospective Cases Undergoing Non-opioid Drug Regimen: Study participants receiving a perioperative non-opioid drug regimen when undergoing unilateral total hip replacement surgery.
  The non-opioid drug regiment includes the following: Guided mindfulness meditation twice daily; Self-administered aromatherapy every 6 hours and at bedtime; Baby aspirin (81mg) twice daily for 6 weeks post surgery; Tylenol/Acetaminophen (1000mg) one pre-operative dose then every 8 hours for three weeks after surgery; Pregabalin twice a day for 2 weeks before surgery and twice a day for 2 weeks after surgery; Prednisone (5mg) Daily for 3 weeks after surgery; Meloxicam (7.5mg) twice a day for 2 weeks before surgery and twice a day, for 2 weeks after surgery; Prilosec (20mg) Daily for 2 weeks before surgery and 2 weeks after surgery; Rescue pain medicine Tramadol (50mg) up to 3 times a day as needed; Voltaren 1% topical arthritis gel up to 4 times daily pre-operative only; Zofran 4 mg pre-operative; Pepcid 20 mg pre-operative; Reglan 10 mg pre-operative; Versed 2 mg pre-operative; Lidocaine (preservative free) height based dosing for subarachnoid block intraoperatively; Propofol 10-125 mcg/kg/min intraoperative; Ancef 2-3 gm weight-based dosing intraoperative; Tranexamic Acid (TXA) 2 gm intraoperative; Decadron 10 mg intraoperative; Local anaesthetic 0.5% bupivacaine hydrochloride intraoperative; Toradol nonsteroidal anti-inflammatory drug max 30 mg intraoperative
- Retrospective Control Underwent Opioid Drug Regimen: A group of retrospective controls that underwent unilateral total hip replacement surgery and used opioid drug regimen perioperatively was initially intended to be created from medical records of patients who had received this surgery in the time prior to this study started, upon conclusion of data collection for the prospective cases. This study did not complete as anticipated and the retrospective control group was not created prior to the early termination of the study.
- Professional Staff: Professional staff who participated in the implementation of the opioid free surgical protocol completed surveys seeking their opinion about interprofessional teamwork and communication.
Period: Overall Study
Arm/Group | Prospective Cases Undergoing Non-opioid Drug Regimen | Retrospective Control Underwent Opioid Drug Regimen | Professional Staff
Started | 7 | 0 | 50
Completed | 6 | 0 | 37
Not Completed | 1 | 0 | 13
Not completed — Withdrawal by Subject | 1 | 0 | 13

BASELINE CHARACTERISTICS:
Population: Baseline information is not available for the retrospective control group as the study was terminated prior to creating this study arm. Only minimal, optional, demographic information was collected from professional staff to maintain anonymity among respondents and to ease their burden of study related activities.
Groups:
- Prospective Cases Undergoing Non-opioid Drug Regimen: Study participants receiving a perioperative non-opioid drug regimen when undergoing unilateral total hip replacement surgery.
- Total: Total of all reporting groups
Arm/Group | Prospective Cases Undergoing Non-opioid Drug Regimen | Retrospective Control Underwent Opioid Drug Regimen | Professional Staff | Total
Number analyzed (Participants) | 7 | 0 | 50 | 57
Age, Categorical [Count of Participants; unit: Participants] — Population: Age was not collected for the professional staff to ensure that survey responses were anonymous.
  Participants
    number analyzed (Participants) | 7 | 0 | 0 | 7
    <=18 years | 0 |  |  | 0
    Between 18 and 65 years | 2 |  |  | 2
    >=65 years | 5 |  |  | 5
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Age was not collected for the professional staff to ensure that survey responses were anonymous.
  years
    number analyzed (Participants) | 7 | 0 | 0 | 7
    (all) | 70 (12) |  |  | 70 (12)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 7 |  | 25 | 32
  Male | 0 |  | 9 | 9
  Other | 0 |  | 3 | 3
  Unknown or not reported | 0 |  | 13 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0 | 0
  Asian | 0 |  | 6 | 6
  Native Hawaiian or Other Pacific Islander | 0 |  | 0 | 0
  Black or African American | 0 |  | 5 | 5
  White | 7 |  | 22 | 29
  More than one race | 0 |  | 0 | 0
  Unknown or Not Reported | 0 |  | 17 | 17
Region of Enrollment [Number; unit: participants]
  United States | 7 |  | 50 | 57

OUTCOME MEASURES:

1. Primary Outcome: Total Post-operative Opioid Requirements With Non-opioid Drug Regimen
Description: Total post-operative opioid requirements (opioid dose) were calculated for participants receiving the non-opioid drug regimen, among participants who required post-operative opioid medication.
Time Frame: Up to 5 weeks
Population: This analysis includes participants who completed the study and required post-operative opioid medication.
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Prospective Cases Undergoing Non-opioid Drug Regimen
Number analyzed (Participants) | 1
milligrams | 400 (0)

2. Secondary Outcome: Nebraska Interprofessional Education Attitude Scale (NIPEAS) Score for Professional Staff Arm
Description: The Nebraska Interprofessional Education Attitude Scale (NIPEAS) was developed to measure the attitudes of pre-clinical learners to practicing health professionals. The NIPEAS is a 19-item questionnaire assessing attitudes related to interprofessional collaboration. Responses were given using a 5-point Likert scale where 1 = Strongly Disagree to 5 = Strongly Agree. The total score is the average of the average scores for each item and ranges from 1 to 5. A higher total score indicates increased positive perceptions toward interprofessional collaboration.
Time Frame: Prior to protocol implementation (baseline), halfway through the recruitment period (2 months) and after the last participant has been discharged from the hospital (4 months)
Population: The baseline survey was provided to all perioperative suite professional staff who gave their consent to participate in the study, however, 13 did not complete the survey. The follow-up surveys were to be completed once the full protocol had been implemented on all 60 anticipated patient participants. As the trial was terminated prior to enrolling 60 participants, the follow-up NIPEAS scale scores were not collected.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Professional Staff
Number analyzed (Participants) | 37
score on a scale
  Baseline | 4.35 (0.39)
  2 months after protocol implementation: number analyzed (Participants) | 0
  4 months after protocol implementation: number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected beginning at the time consent to participate in the study was given, up 5 weeks post-surgery for patient participants, or upon completion of the baseline survey for professional staff participants.
Description: Information on adverse events is not available for the retrospective control group as the study was terminated prior to creating this study arm.
Arm/Group | Prospective Cases Undergoing Non-opioid Drug Regimen | Professional Staff
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/37
Other Adverse Events (participants affected / at risk) | 0/7 | 0/37

LIMITATIONS AND CAVEATS:
This study aimed to enroll a total of 170 participants. Due to staffing issues and the coronavirus disease 2019 (COVID-19) pandemic, this trial was terminated early and therefore the retrospective data was not collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-08): https://cdn.clinicaltrials.gov/large-docs/96/NCT04766996/Prot_SAP_000.pdf